CLINICAL TRIAL: NCT01675804
Title: A Randomized Clinical Trial Comparing Computer-assisted Cognitive Rehabilitation (CACR), Psycho-stimulants, and Placebo CACR in the Treatment of Attention Deficit/ Hyperactivity Disorder
Brief Title: Computer-assisted Cognitive Rehabilitation (CACR), Placebo CACR and Psycho-stimulants in the Treatment of ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allameh Tabatabai University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 83-6516
Record Dates: First submitted 2012-07-29; First posted 2012-08-30 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Computerized cognitive rehabilitation (Experimental): -Computer-assisted cognitive rehabilitation (CACR): 20 Ninety-minute sessions of CACR.
  Interventions: Other: Computerized cognitive rehabilitation
- Placebo CACR [PCACR] (Placebo Comparator): -PCACR group simultaneously received 20 Ninety-minute sessions of Placebo CACR.
  Interventions: Other: Placebo CACR [PCACR]
- Ritalin (Experimental): -2 to 3 doses of 10 mg Ritalin tablets per day during two months.
  Interventions: Drug: Ritalin

INTERVENTIONS:
Other: Computerized cognitive rehabilitation — - Computerized cognitive rehabilitation: 20 ninety-minute sessions of computerized cognitive rehabilitation.
  Arms: Computerized cognitive rehabilitation
Drug: Ritalin — -drug therapy: 2 or 3 doses of 10 mg tablets of Immediate-release Methylphenidate (Ritalin) per day for 2 months.
  Other Names: Immediate release methylphenidate
  Arms: Ritalin
Other: Placebo CACR [PCACR] — PCACR: 20 ninety-minute sessions of Placebo computerized cognitive training.
  Arms: Placebo CACR [PCACR]

SUMMARY:
Current research aimed to compare the efficacy of computer-assisted cognitive rehabilitation (CACR), stimulant drugs and Placebo CACR on executive functions and clinical symptoms of children with attention deficit/hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
The investigators administered a randomized controlled trial (RCT) through random assignment of ADHD subjects in to three different groups to compare the effects of CACR, immediate-release methylphenidate, and a Placebo CACR (i.e. some computerized tasks assumed not having any therapeutic effects) on the functioning of children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosis
* age between 7 and 12
* IQ > 85

Exclusion Criteria:

* sever co-morbid disorder
* seizure
* IQ < 85
* disability
* sever medical condition

Ages: 7 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Persian software for the continuous performance test [CPT] | 5 months
  The Persian software of CPT is a visual CPT test.
Persian software for the Tower of London Test [TOL] | 5 months
  Persian TOL is a software version of tower of London test (TOL) which was developed in Iran.
Forward/Reversed digit span tasks from the WISC-R testing battery. | 5 months
  Reversed digit span from the WISC-R (Wechsler, 1974) was used to measure executive verbal WM and the forward digit span was used to measure short-term memory.
Raven's colored progressive matrices. | 5 months
  Raven's colored progressive matrices (Raven, 1995) was used to measure complex non-verbal reasoning.
Span board task from the Lumosity.com online software (Lumosity.com, 2012) | 5 months
SNAP-IV scales | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Saeed Azami, MSc, Principal Investigator — Candidate for PhD in Psychology, Department of Psychology, Semnan University, Semnan, Iran; Alireza Moghadas, PhD, Study Director — Department of Clinical Psychology, Allameh Tabatabaei University, Tehran, Iran.; Faramarz Sohrabi, PhD, Study Director — Department of Clinical Psychology, Allameh Tabatabaei University, Tehran, Iran.; Morteza Nazifi, PhD, Study Director — Department of psychology, University of Bojnord, Bojnord, Iran.
Locations (1):
- Counseling and guidence Center of the Department of education of region 9 of Tehran, Tehran, Tehran Province, Iran